CLINICAL TRIAL: NCT04130321
Title: Demonstration of the Prebiotic-like Effects of Camu-camu Consumption Against Obesity-related Disorders in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, André Marette, Professor, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CAMU 2020-3350
Record Dates: First submitted 2019-10-03; First posted 2019-10-17 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Overweight; Microtia; Endotoxemia; Metabolic Syndrome; Insulin Resistance; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Overweight; Congenital Microtia; Endotoxemia; Metabolic Syndrome; Insulin Resistance; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Camu camu (Experimental)
  Interventions: Dietary Supplement: Camu camu
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Camu camu — 3 capsules of camu camu powder (500 mg / capsule) daily during 12 weeks
  Arms: Camu camu
Dietary Supplement: Placebo — 3 capsules of placebo daily during 12 weeks
  Arms: Placebo

SUMMARY:
Previous work of the investigators demonstrated the anti-obesity and anti-steatosis potential of the Amazonian fruit camu-camu (CC) in a mouse model of diet-induced obesity [1]. It was demonstrated that the prebiotic role of CC was directly linked to higher energy expenditure stimulated by the fruit since fecal transplantation from CC-treated mice to germ-free mice was sufficient to reproduce the effects.

The full protection against hepatic steatosis observed in CC-treated mice is of particular importance since nonalcoholic fatty liver disease (NAFLD) is one of the most common causes of chronic liver disease. Thirty percent of adults in developed countries have excess fat accumulation in the liver, and this figure can be as high as 80% in obese subjects. NAFLD is an umbrella term encompassing simple steatosis, as well as non-alcoholic steatohepatitis which can lead to cirrhosis and hepatocellular carcinoma in up to 20% of cases. Up to now, except for lifestyle changes, no effective drug treatment are available. Previous work has suggested that CC possesses anti-inflammatory properties and could acutely reduce blood pressure and glycemia after a single intake. While CC could represent a promising treatment for obesity and fatty liver, no studies have thoroughly tested this potential in humans. Therefore, a robust clinical proof of concept study is needed to provide convincing evidence for a microbiome-based therapeutic strategy to counteract obesity and its associated metabolic disorders.

The mechanism of action of CC could involve bile acid (BA) metabolism. BA are produced in the liver and metabolized in the intestine by the gut microbiota. Conversely, they can modulate gut microbial composition. BA and particularly, primary BA, are powerful regulators of metabolism. Indeed, mice treated orally with the primary BA α, β muricholic (αMCA, βMCA) and cholic acids (CA) were protected from diet-induced obesity and hepatic lipid accumulation. Interestingly, the investigators reported that administration of CC to mice increased the levels of αMCA, βMCA and CA. Primary BA are predominantly secreted conjugated to amino acids and that deconjugation rely on the microbial enzymatic machinery of gut commensals. The increased presence of the deconjugated primary BA in CC-treated mice indicate that a cluster of microbes selected by CC influence the BA pool composition. These data therefore point to an Interplay between BA and gut microbiota mediating the health effects of CC.

Polyphenols and in particular procyanidins and ellagitannins in CC can also be responsible for the modulation of BA that can impact on the gut microbiota. Indeed, it has been reported that ellagitannins containing food like walnuts modulate secondary BA in humans whereas procyanidins can interact with farnesoid X receptors and alter BA recirculation to reduce hypertriglyceridemia. These effects are likely mediated by the remodeling of the microbiota by the polyphenols.

In accordance with the hypothesis that the ultimate effect of CC is directly linked to a modification of the microbiota, fecal transplantation from CC-treated mice to germ-free mice was sufficient to recapitulate the lower weight gain and the higher energy expenditure seen in donor mice.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 40 kg/m2
* Fasting triglyceride > 1,35 mmol/L
* Understanding of spoken and written french
* Accept to follow study instructions

Exclusion Criteria:

* Smoking
* Medication affecting glucose metabolism, blood lipid levels or blood pressure
* Metabolic disorders requiring treatment
* Diabetic subjects presenting HbA1c >6.5% or fasting glycemia >7 mmol/L
* Consumption of fruit or polyphenol supplements in the last 3 months
* Allergy or intolerance for camu camu or for an ingredient of the placebo
* Alcohol consumption of > 2 drinks / day
* Weight change > 5% of body weight in the last 3 months
* Major surgical operation in the last 3 months or planned in the next months
* Pregnant or breastfeeding women or women planning pregnancy in the next months
* Antibiotics intake in the last 3 months
* Regular probiotics intake in the last 3 months
* Gastrointestinal malabsorption
* Cirrhosis
* Chronic kidney disease
* Concomitant participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-10-31 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Change in Gut Microbiota Composition and Diversity | Change between the beginning and the end of each treatment (12 weeks each)
  Global variation of the fecal microbiota
Change in fat accumulation in the liver | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of fat accumulation by magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Change in Endotoxemia | Change between the beginning and the end of each treatment (12 weeks each)
  Plasma Lipopolysaccharides (LPS) and Lipopolysaccharide Binding Protein (LBP)
Change in Intestinal permeability | Change between the beginning and the end of each treatment (12 weeks each)
  Plasma zonulin
Change in Inflammation state of the tissue | Change between the beginning and the end of each treatment (12 weeks each)
  Fecal calprotectin and chromogranin
Change in Short chain and branched chain fatty acids in the feces | Change between the beginning and the end of each treatment (12 weeks each)
  Measure short chain fatty acids in the feces
Change in gut health | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of gastrointestinal symptoms using a standardized questionnaire (the gastrointestinal symptom rating scale (GSRS))
Change in stool consistency | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of stool consistency using a standardized questionnaire (Bristol stool chart)
Change in Glucose homeostasis | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of plasma glucose using a 3-hour oral glucose tolerance test
Change in Glucose homeostasis | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of insulin concentration using a 3-hour oral glucose tolerance test
Change in Glucose homeostasis | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of c-peptide concentration using a 3-hour oral glucose tolerance test
Change in Glucose homeostasis | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of glycated haemoglobin
Change in Lipid profile | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of plasma triglycerides (TG), Total cholesterol, LDL, HDL, Apolipoprotein B and free fatty acids
Change in anthropometric measurements | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of BMI (measured with weight change and height throughout the protocol)
Change in anthropometric measurements | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of waist circumference
Change in body composition | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of body composition by osteodensitometry
Change in chronic inflammation | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of plasma high sensitive C-Reactive Protein (hs-CRP)
Change in liver health | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of aspartate transaminase and alanine aminotransferase (AST and ALT)
Change in gene expression levels | Change between the beginning and the end of each treatment (12 weeks each)
  Transcriptomic analyses to investigate underlying mechanisms of action
Change in circulating levels of plasma metabolites | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of camu-camu derived metabolites, short chain fatty acids, branched chain fatty acids, bile acids, phenolic compounds
Change in camu camu-derived metabolites present in stool | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of metabolome: camu-camu derived metabolites, short chain fatty acids, branched chain fatty acids, bile acids, phenolic compounds
Change in blood pressure | Change between the beginning and the end of each treatment (12 weeks each)
  Evaluation of systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- INAF, Université Laval, Québec, Canada